CLINICAL TRIAL: NCT01712347
Title: An Open-Label, Multicenter, Non-Interventional, Observational Study To Assess The Effect Of First Line Bevacizumab Treatment With Fluoropyrimidine-Based Chemotherapy (CTX) In Patients With Metastatic Colorectal Cancer
Brief Title: An Observational Study of First-Line Bevacizumab (Avastin) With Fluoropyrimidine-Based Chemotherapy in Participants With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28233
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mCRC Participants: mCRC participant will receive bevacizumab as per approved label with the approved first-line fluoropyrimidine based chemotherapy, as per physician discretion. The protocol does not specify the chemotherapy regimen to be used, the choice of chemotherapy will be at the discretion of treating physician.
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered as per approved label.
  Other Names: Avastin
Drug: Chemotherapy — The protocol does not specify the chemotherapy regimen to be used, the choice of chemotherapy will be at the discretion of treating physician.

SUMMARY:
This multicenter observational study will evaluate the efficacy and safety of first-line bevacizumab (Avastin) in combination with fluoropyrimidine-based chemotherapy in participants with metastatic colorectal cancer (mCRC). Participants for whom the treating physician has decided to initiate first-line fluoropyrimidine based chemotherapy in combination with bevacizumab will be observed for approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed metastatic colorectal cancer who will receive bevacizumab in combination with first-line fluoropyrimidine-based chemotherapy

Exclusion Criteria:

* Participants not qualified for bevacizumab treatment according to the local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic colorectal cancer receiving first-line bevacizumab in combination with fluoropyrimidine-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival from the time of starting first-line therapy | Start of first line therapy until death (up to approximately 4 years)

SECONDARY OUTCOMES:
Progression-free survival from the time of starting first-line therapy, assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria | Start of first line therapy until death (up to approximately 4 years)
Percentage of participants with best overall response, assessed according to RECIST v.1.1 criteria | Start of first line therapy until death (up to approximately 4 years)
Percentage of participants with liver resection | up to approximately 4 years
Number of participants with adverse events | up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Taiwan (9):
  - Chang Gung Medical Foundation - Chai Yi; Surgery, CHAI YI
  - Kaohsiung Chang Gung Memorial Hospital; Colorectal Surgery, Kaohsiung City
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - Taichung Veterans General Hospital; Dept of Surgery, Taichung
  - National Cheng Kung Uni Hospital; Dept of Hematology and Oncology, Tainan
  - Veterans General Hospital; Division of Oncology, Taipei
  - Tri-Service General Hospital; Hematology and Oncology, Taipei
  - Mackay Memorial Hospital; Department of Surgery, Division of Colon and Rectal Surgery, Taipei
  - Chang Gung Medical Foundation - Linkou; Colo-rectal Surgery, Taoyuan District